CLINICAL TRIAL: NCT05354609
Title: Assessment of Intestinal Inflammatory Activity in the Follow-up of Patients With Crohn's Disease: Diffusion-weighted MR-enterography, Without or With Bowel Cleansing, Compared With Standard MR-enterography
Brief Title: DWI MR-enterography Without or With Bowel Cleansing to Assess Intestinal Inflammatory Activity in the Follow-up of Crohn's Disease
Acronym: ENTEDIF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2022_843_0013
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease; Bowel Cleansing; Apparent Diffusion Coefficient
Keywords: Crohn Disease; diffusion-weighted imaging; MR-enterography; bowel cleansing; apparent diffusion coefficient
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-enterography (Experimental)
  Interventions: Other: MR-enterography

INTERVENTIONS:
Other: MR-enterography — All patients will undergo a simplified MR-enterography, which includes four sequences, without bowel cleansing or injection. On the same day, the standard MR-enterography will be performed as in clinical practice, after ingestion of the usual oral preparation.

SUMMARY:
Since 2009, many studies tend to prove the effectiveness of diffusion-weighted MR-enterography in the assessment of inflammatory activity in IBD compared to standard MR-enterography, with the emergence of new radiological scores such as the Clermont score. Diffusion-weighted MRI (DWI) is a faster technique and does not require the injection of gadoline contrast medium, which is a desirable in view of recent data on their long-term adverse effects (intracerebral deposits, nephrogenic systemic fibrosis).

The advent of 3T MRI, which provides a better signal, a better spatial resolution or the same examination quality in a shorter time, seems promising for the future of DWI.

However, to date, there are still few studies carried out at 3T in this field or even few studies on the possibility of doing away with bowel cleansing, although this is one of the main demands of patients. All patients will undergo a simplified MR-enterography, which includes four sequences, without bowel cleansing or injection. On the same day, the standard MR-enterography will be performed as in clinical practice, after ingestion of the usual oral preparation.

Three reading sessions of the examination will be organized at intervals of at least one month by two radiologists specialized in digestive imaging, blinded to the clinical and

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with Crohn's disease with bowel involvement for whom a MR-enterography was ordered as part of their follow-up
* Age ≥ 18
* Subject's ability to understand and express opposition
* Affiliation to French social security system

Exclusion Criteria:

* Any contraindication to MRI
* Allergy to gadolinium chelates
* Claustrophobia
* Major obesity that does not allow the patient to enter the machine's tunnel (whose diameter is 70 cm)
* Pregnant woman
* Person under curators or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
variation of inflammatory activity localisation number in the main bowel | one day
  variation of inflammatory activity localisation number in the main bowel between diffusion entero-MRI with bowel cleansing versus standard enteroMRI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No